CLINICAL TRIAL: NCT05364112
Title: Utilization of Compreflex Wraps in Patients With Chronic Venous Insufficiency: A Quasiexperimental Post-market Clinical Follow-up Study
Brief Title: Utilization of Compreflex Wraps in Patients With Chronic Venous Insuffciency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuala Lumpur General Hospital (Other Government)
Collaborators: SULTAN AHMAD SHAH MEDICAL CENTRE @ IIUM (Unknown); Universiti Kebangsaan Malaysia Medical Centre (Other); University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Harikrishna K.Ragavan Nair, Head of Wound Care Unit, Department of Medicine, Kuala Lumpur General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-21-330-58451
Record Dates: First submitted 2022-05-01; First posted 2022-05-06 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Varicose Ulcer; Venous Insufficiency of Leg
Keywords: Varicose Ulcer; Compression Bandages; Venous Insufficiency of Leg; Stockings, Compression
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compreflex (Experimental): Patients recruited for the study will be given one unit of Compreflex (study device) to be worn on the studied leg with a venous ulcer. Once the wound is covered by dressing, the subjects were instructed to wear the study device for 24 hours over the study period. Subjects were allowed to take off the study device during a shower. Subjects were asked to visit the clinic for follow-up purposes at 3 assessment time points after being recruited at the first visit: V2 (3-week), V3 (12-week) and V4 (26-week). Subjects' wound area, leg circumferences were measured and calculated. Patient-centred questionnaires were given to the subjects to assess their compliance and satisfaction with the study device.
  Interventions: Device: Compreflex

INTERVENTIONS:
Device: Compreflex — The Compreflex standard calf and foot (with basic liner) from Sigvaris (St. Gallen, Switzerland) is an easy-to-use interlacing Velcro wrap device with adjustable compression levels.

SUMMARY:
This is a multicentre, quasi-experimental study to evaluate the Conformitè Europëenne-marked Compreflex standard calf and foot (with basic liner) under routine conditions.

The study will be conducted at 4 clinics and will include 100 consecutive patients. Patients will be followed-up until 26 weeks.

DETAILED DESCRIPTION:
In chronic venous insufficiency (CVI), the venous system of the legs is ineffective in performing venous return, and there is venous reflux due to valve failure, physical inactivity and cardiovascular problems, leading to an increase in the pressure in the veins and venous hypertension. Chronic venous insufficiency includes a range of signs and symptoms, including varicose veins, varicose veins, oedema, skin lesions and ulcers.

Venous ulcers are wounds that occur due to improper functioning of venous valves secondary to severe chronic venous insufficiency. They are mainly located in the internal lateral zone of the distal third of the leg. Ulcers of venous aetiology make up 80% of all ulcers. They have an incidence of between 15 to 30 per 100'000 personyears.

The median healing time for chronic venous ulcers approximates 180 days. These ulcers may produce a foul-smelling discharge, can become infected and cause pain, which, in combination with slow healing and frequent relapses, affects the quality of life of affected patients.

The treatment of chronic venous ulcers requires a comprehensive approach for the patient, addressing the etiological factors that determine their evolution, such as venous insufficiency, diet, physical inactivity and postural measures. Local treatment has two components: local ulcer healing and control of venous insufficiency by means of compression therapy.

There is evidence that compression therapy promotes the healing process of venous ulcers. However, there is a large number of compression garments available and it is unclear which method of compression is the most effective. Traditionally, multilayered compression banding was the first line management for uncomplicated venous ulcers. This serves to increase venous return and reduce venous hypertension, as well as reduce oedema and improve lymphatic circulation. Despite its importance and widespread use, it has been reported that ca. 50% of patients do not comply with their multilevel bandaging. Reasons for non-compliance are skin irritation, bandage slippage, pain, malodor, inability to maintain hygiene, and discomfort and inability to wear normal footwear. Over recent years, there has been development of several Velcro-based wrap devices for use as alternative compression bandaging for venous ulcer management, using either interlacing or overlapping technique of wrapping. Systematic reviews have been undertaken for Velcro wrap devices, including their use in chronic edema, lipedema, and lymphedema, as well as venous ulceration. These systematic reviews were able to show a reduction in limb volume and more consistent sub-bandage pressure in Velcro wrap devices compared with bandaging. In addition, one of the major advantages that was reported was the relative ease to remove and reapply these devices, which can, therefore, encourage self-care, improve independence and, potentially, quality of life.

The Compreflex standard calf and foot (with basic liner) from Sigvaris (St. Gallen, Switzerland) is an easy to use interlacing Velcro wrap device with adjustable compression levels.This Compreflex wrap is intended for patients with mild to moderate lymphedema and venous insufficiency. More than 200'000 products have been sold worldwide since 2016. The product is being used in many European countries (including United Kingdom, Switzerland, Netherland), United States of America, Saudi Arabia, India, Indonesia, Taiwan and Hong Kong, with no product-related safety issues reported. Although the product is not substantially different from other established products that are already available on the market, there are no clinical data published on Compreflex.

The present study was therefore designed to confirm the performance of the Compreflex standard calf and foot (with basic liner).

ELIGIBILITY:
Inclusion Criteria:

* Are patients for whom it is medically indicated to use the device of interest in accordance with its instruction for use
* Are between 18 and 80 years old
* Have provided informed consent
* Are willing and able to participate in the follow-up examinations

Exclusion Criteria:

* Lymphoedema
* Presence of other comorbidities (i.e. congestive cardiac failure, renal failure, fulminant hepatic failure)
* Pregnancy
* Septicemia
* Infected chronic venous ulcer wound
* Ischemia (ABSI<0.8)
* Noncompressible arteries (ABSI<0.8)
* Bleeding tendencies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound size | 26 months
  Ulcer size will be measured by Measuring the length "head-to-toe" at the longest point. Measure the width side-to-side at the widest point that is perpendicular to the length.
  The inner border of the wound will be used for reference, both for length and width.

SECONDARY OUTCOMES:
Oedema volume | 26 months
  Limb circumference measurement will be performed as indicated in the figure below, with:
  00: level of ground; 0: tip of great toe; C1: base of metatarsophalangeal joints; C2: 10 cm from 0; C3: midtarsal line through most proximal part of dorsum of foot; C4: line through midpoint of lateral malleolus; C5: 12 cm from 00; C6: 20 cm from 00; C7: 30 cm from 00; L1: length from 0 to C3; L2: length from 00 to C4; L3: length from C4 to C7.
  Volume of edema will then be estimated as follows:

CONTACTS AND LOCATIONS:
Overall Officials: Harikrishna R Nair, Principal Investigator — Kuala Lumpur General Hospital
Locations (1):
- Wound Care Unit, Dept. of Internal Medicine, Kuala Lumpur Hospital, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No